CLINICAL TRIAL: NCT06791070
Title: A Prospective Multicenter Clinical Trial on the Efficacy and Safety of RC48-ADC (Disitamab Vedotin) Combined With Toripalimab in Advanced HER2-positive Extramammary Paget Disease of the Scrotum
Brief Title: A Study of RC48-ADC Combined With JS001 for Advanced Extramammary Paget Disease of the Scrotum
Acronym: RC48&J for EPD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Collaborators: Zhejiang Tumor Hospital (Other); Fujian Provincial Hospital (Other); Zhangzhou Affiliated Hospital of Fujian Medical University (Other); Quanzhou First Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024YF066-01; ECCO-KY-24003 (Other Grant/Funding Number: Eastern Clinical Oncology Research Center)
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Paget Disease, Extramammary; Scrotum Disease
Keywords: extramammary Paget disease; Disitamab Vedotin; Toripalimab; RC48-ADC
MeSH Terms: conditions — Paget Disease, Extramammary | interventions — toripalimab

STUDY DESIGN:
Intervention Model Description: Multiple center, single arm, open label, prospective phase II study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Disitamab Vedotin combined with Toripalimab
  Interventions: Drug: Disitamab Vedotin combined with Toripalimab

INTERVENTIONS:
Drug: Disitamab Vedotin combined with Toripalimab — Disitamab Vedotin at a dosage of 2mg/kg and 3mg/kg of Toripalimab administered intravenously every 3 weeks (ivgtt q3w) is continued until disease progression, with the allowance for treatment discontinuation due to disease progression, death, intolerable toxicity, withdrawal of informed consent, initiation of new antineoplastic therapy, or other reasons specified in the protocol, with the earliest occurring event taking precedence. Alternatively, the study investigator may determine the need to discontinue treatment.

SUMMARY:
The goal of this clinical trial is to learn if Disitamab Vedotin combined with Toripalimab works to treat advanced HER2-positive extramammary Paget disease of the scrotum. It will also learn about the safety of this combination. The main questions it aims to answer are: Does this combination reduce tumor volume and delay disease progression? What medical problems do participants have when receving this combination? Participants will: Intravenous using this combination every 3 weeks until disease progression or intolerable adverse reactions occur. Visit the clinic once every 3 weeks for checkups and tests.

DETAILED DESCRIPTION:
This study is a multiple-center, phase II clinical trial. Participants with HER2-positive advanced scrotal extramammary Paget's disease who met the eligibility criteria were enrolled after signing an informed consent form. All patients received treatment with 2mg/kg of Disitamab Vedotin and 3mg/kg of Toripalimab intravenous infusion every 3 weeks until disease progression. Follow-up was conducted until disease progression, intolerable adverse reactions, withdrawal of informed consent by the participant, loss to follow-up, or death. The area of the largest lesion on the scrotal skin was measured and clinical tumor imaging assessments were performed using RECIST during the treatment process.

ELIGIBILITY:
Inclusion Criteria:

Voluntarily sign the informed consent form and comply with the requirements of the protocol.

Age ≥ 18 years old. Confirmed diagnosis by histological examination, combined with imaging assessment for scrotal extramammary Paget's disease; pathologically confirmed as HER2 positive, i.e., immunohistochemical test HER2 ≥ 1+.

ECOG score: 0 to 1. At least one measurable lesion (according to the RECIST criteria, non-nodal lesions with a longest diameter on CT scan ≥10 mm, and nodal lesions with a shortest diameter on CT scan ≥15 mm); or skin lesions that can be evaluated according to the WHO criteria.

Adequate organ function: Blood routine: Absolute Neutrophil Count (ANC) ≥1.5×10^9/L, Platelet (PLT) ≥70×10^9/L, Hemoglobin (HGB) ≥80g/L; Liver function: Total Bilirubin (TBIL) ≤1.5×Upper Limit of Normal Value (ULN); Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤3×ULN; Serum Albumin ≥28 g/L; Alkaline Phosphatase (ALP) ≤5×ULN; If the subject has received routine liver protection treatment and meets the above standards, and is stable for at least one week after assessment by the researcher, they may be enrolled; Renal function: Serum Creatinine (Cr) ≤1.5×ULN, or Creatinine Clearance ≥50 mL/min (using the standard Cockcroft-Gault formula): Coagulation function: International Normalized Ratio (INR) ≤1.5 / Prothrombin Time (PT) ≤1.5×ULN, Activated Partial Thromboplastin Time (aPTT) ≤1.5×ULN; If the subject is receiving anticoagulant therapy, as long as PT and INR are within the range specified for the anticoagulant medication, it is acceptable.

Estimated life expectancy ≥3 months.

Exclusion Criteria:

Have a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation; Have had active autoimmune diseases within 2 years prior to the start of the study treatment that required systemic treatment (such as the use of disease-modifying drugs, corticosteroids, or immunosuppressants), except for replacement therapies (e.g., thyroid hormone, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency); currently receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy. The dose is >10mg/day of prednisone or other equivalent hormones, and it is within 2 weeks of the first administration and still in use; Have a history of active tuberculosis; Have uncontrollable, recurrent drainage of ascites, pericardial effusion, or pleural effusion; Have undergone major organ transplantation; Received major surgical treatment, incisional biopsy, or significant traumatic injury within 28 days prior to the start of the study treatment; or have chronic non-healing wounds or fractures; Have a history of live attenuated vaccine administration within 14 days prior to the start of the study treatment or plan to receive live attenuated vaccine vaccination during the study period; Have had a severe hypersensitivity reaction after the use of monoclonal antibodies; known allergy to the active ingredients or excipients of this study drug; Within 4 weeks prior to the start of the study, are participating in or have participated in other clinical studies; Have a history of severe allergies; Have a risk of bleeding, or coagulation dysfunction, or are currently receiving -thrombolytic therapy; Have a history of substance abuse and are unable to quit or have mental disorders; According to the investigator's judgment, there are concomitant diseases that seriously endanger the safety of the subject or affect the completion of the study, or there are other reasons deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | every 6 weeks,up to 24 weeks
  ORR includes two categories:
  Complete Response (CR): All target lesions in the patient have completely disappeared, and no new lesions have appeared for a certain time.
  Partial Response (PR): The tumor in the patient has reduced in size by at least 30%, and this reduction has been maintained for a certain period.

SECONDARY OUTCOMES:
Progression free survival | through study completion, an average of 2 year
  Progression-Free Survival (PFS) is a clinical endpoint used primarily in oncology to measure the effectiveness of a treatment in delaying the progression of a disease. It is defined as the length of time during which a patient's disease does not get worse after starting a treatment. PFS takes into account the time from the start of treatment until the first occurrence of disease progression, or the patient's death if it occurs before progression.
Adverse events | through study completion, an average of 2 year
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Shaoxing Zhu, Doctor, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data is protected.

REFERENCES:
- See also: Related Info — https://www.chictr.org.cn/